CLINICAL TRIAL: NCT01833728
Title: A Comparison of Nefopam-propacetamol Combination and Propacetamol for Postoperative Quality of Recovery After Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0023
Record Dates: First submitted 2013-04-14; First posted 2013-04-17 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Renal Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — propacetamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- nefopam-propacetamol combination group (Experimental)
  Interventions: Drug: nefopam-propacetamol combination
- propacetamol alone group (Active Comparator)
  Interventions: Drug: propacetamol alone

INTERVENTIONS:
Drug: nefopam-propacetamol combination — Patients in both groups will receive intravenous patient-controlled analgesia (PCA) using fentanyl.
  In nefopam-propacetamol combination group, patients will receive nefopam(20mg mixed to normal saline 100mL) and propacetamol(2g mixed to normal saline 100mL), 30 minutes before the end of operation, every 6 hours for up to 48 hours.
  Arms: nefopam-propacetamol combination group
Drug: propacetamol alone — In propacetamol alone group, patients will receive placebo (normal saline 2 ml mixed to normal saline 100mL) and propacetamol(2g mixed to normal saline 100mL), 30 minutes before the end of operation, every 6 hours for up to 48 hours.
  Arms: propacetamol alone group

SUMMARY:
The multimodal analgesia for postoperative pain aims for optimal analgesia through additive or synergic drug effects. The multimodal analgesia results in the use of smaller doses of opioids and lowering opioid-related side effects.

Non-opioid analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), propacetamol (prodrug of acetaminophen), nefopam are often given along with opioids as part of multimodal analgesia after major surgery.

NSAIDS, commonly used non-opioid analgesics, have gastro-intestinal, renal, and cardiac side effects.

In contrast, propacetamol or nefopam, two drugs with central analgesic effects, can be safely used as analgesic adjuvants with opioid after nephrectomy, because these drugs do not alter renal function or cause hemorrhagic complications.

Recent study demonstrated that the antinociceptive properties of paracetamol (intravenous acetaminophen) associated with the analgesic effectiveness of nefopam could explain the observed synergy of the combination.

The aim of this randomized, double-blinded study is to compare the opioid-sparing effect and analgesic efficacy, as well as quality of recovery, of nefopam-propacetamol combination and propacetamol in patients undergoing laparoscopic nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1-3,
* aged 20 to 65 years,
* undergoing laparoscopic nephrectomy

Exclusion Criteria:

* Severe cardiac disease,
* hepatic insufficiency,
* chronic kidney disease stage ≥3,
* preoperative use of analgesics(corticosteroids, opioid),
* chronic alcoholics,
* hemolytic anemia,
* convulsions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | at 24 hours postoperative
  Quality of recovery questionnaire score at 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative opioid consumption | at 24 and at 48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Mimoz O, Incagnoli P, Josse C, Gillon MC, Kuhlman L, Mirand A, Soilleux H, Fletcher D. Analgesic efficacy and safety of nefopam vs. propacetamol following hepatic resection. Anaesthesia. 2001 Jun;56(6):520-5. doi: 10.1046/j.1365-2044.2001.01980.x. PMID 11412156
- [Background] Girard P, Niedergang B, Pansart Y, Coppe MC, Verleye M. Systematic evaluation of the nefopam-paracetamol combination in rodent models of antinociception. Clin Exp Pharmacol Physiol. 2011 Mar;38(3):170-8. doi: 10.1111/j.1440-1681.2011.05477.x. PMID 21226753